CLINICAL TRIAL: NCT01369849
Title: Phase I/II Study of the Combination of Bendamustine, Rituximab and MK-2206 in the Treatment of Relapsed Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Brief Title: Akt Inhibitor MK2206, Bendamustine Hydrochloride, and Rituximab in Treating Patients With Relapsed Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02675; NCI-2011-02675 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000701372; NCCTG-N1087; N1087 (Other: Alliance for Clinical Trials in Oncology); N1087 (Other: CTEP); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — MK 2206; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Akt inhibitor MK2206, bendamustine, rituximab) (Experimental): Patients receive Akt inhibitor MK2206 PO on days 1, 8, 15, and 22 (days 1, 8, 15, 22, and 29 of course 1); rituximab IV on day 1 (day 8 of course 1); and bendamustine hydrochloride IV over 30-60 minutes on days 1-2 (days 8-9 of course 1). Treatment repeats every 28 days (35 days for course 1 and 84 days for course 6) for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Bendamustine Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Rituximab

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Bendamustin Hydrochloride; Cytostasan Hydrochloride; Ribomustin; SyB L-0501; Treanda
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83

SUMMARY:
This phase I/II trial studies the side effects and best dose of v-akt murine thymoma viral oncogene homolog 1 (Akt) inhibitor MK2206 when given together with bendamustine hydrochloride and rituximab and to see how well they work in treating patients with refractory chronic lymphocytic leukemia or small lymphocytic lymphoma. Akt inhibitor MK2206 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving Akt inhibitor MK2206 with bendamustine hydrochloride and rituximab may be an effective treatment for relapsed chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and maximum tolerated dose (MTD) of MK-2206 (Akt inhibitor MK2206) in combination therapy with bendamustine (bendamustine hydrochloride)-rituximab in relapsed chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) patients. (Phase I) II. To assess the rate of complete response (CR) of MK-2206 in combination with bendamustine-rituximab in relapsed CLL or SLL patients. (Phase II)

SECONDARY OBJECTIVES:

I. To assess clinical efficacy of MK-2206 in combination with bendamustine-rituximab as demonstrated by analysis of overall response rate (CR, complete response with incomplete bone marrow recovery [CRi], clinical complete response [CCR], near partial response [nPR] and partial response [PR]), duration of response, and treatment free survival.

II. To assess the toxicity profile of MK-2206 in combination with bendamustine-rituximab.

TERTIARY OBJECTIVES:

I. Evaluation of whether the established CLL prognostic factors (cluster of differentiation [CD]38, CD49d, immunoglobulin heavy chain variable [IGHV], fluorescence in situ hybridization [FISH] and zeta-chain-associated protein kinase 70 [ZAP-70]) predict responses to the combination therapy of MK2206, with bendamustine-rituximab.

II. Minimal residual disease will be evaluated after treatment in patients who achieve a clinical response; minimal residual disease (MRD) status will be explored in relation to both the quality and duration of response.

III. Evaluation of the effects of the addition of MK-2206 to bendamustine-rituximab on B cell receptor initiated, phosphoinositide 3-kinase (PI3K)/Akt downstream signal pathways, apoptosis analysis and leukemic cell activation status, as well as multiple cytokine profiles and key gene expression analysis with focus on leukemic cells.

IV. Evaluation of marrow stromal cells (MSC)-CLL biology including the effects of the addition of MK-2206 to bendamustine-rituximab on CLL marrow stromal cell (MSC) proliferation, migration and cytokine production, as well as the adhesion capacity between MSC and leukemic cells.

OUTLINE: This is a phase I, dose-escalation study of Akt inhibitor MK2206 followed by a phase II study.

Patients receive Akt inhibitor MK2206 orally (PO) on days 1, 8, 15, and 22 (days 1, 8, 15, 22, and 29 of course 1); rituximab intravenously (IV) on day 1 (day 8 of course 1); and bendamustine hydrochloride IV over 30-60 minutes on days 1-2 (days 8-9 of course 1). Treatment repeats every 28 days (35 days for course 1 and 84 days for course 6) for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 or 12 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) according to the National Cancer Institute (NCI) criteria or small lymphocytic lymphoma (SLL) according to the World Health Organization (WHO) criteria; this includes previous documentation of:

  * Biopsy-proven SLL or
  * Diagnosis of CLL according to NCI working group criteria as evidenced by all of the following:

    * Peripheral blood B-cell count of > 5 x 10^9/L consisting of small to moderate size lymphocytes
    * Immunophenotyping consistent with CLL defined as:

      * The predominant population of lymphocytes share both B-cell antigens (CD19, CD20 [typically dim expression], or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3,CD2, etc.)
      * Clonality as evidenced by kappa (Κ) or lambda (λ) light chain expression (typically dim immunoglobulin expression) or other genetic method (e.g., immunoglobulin heavy chain variable [IGHV] analysis)
      * NOTE: splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
    * Before diagnosing CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative fluorescence in situ hybridization (FISH) analysis for t (11;14) (IgH/CCND1) on peripheral blood or tissue biopsy, or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy
* Demonstrated progression after one or two prior lines of CLL therapy; note: rituximab monotherapy does not count as a prior line of therapy
* Progressive disease with any one of the following characteristics based on standard criteria for treatment as defined by the NCI-Working Group (WG) 1996

  * Symptomatic CLL characterized by any one of the following:

    * Weight loss >= 10% within the previous 6 months
    * Extreme fatigue attributed to CLL
    * Fevers > 100.5° Fahrenheit (F) for 2 weeks without evidence of infection
    * Drenching night sweats without evidence of infection
  * Evidence of progressive bone marrow failure with hemoglobin < 11 g/dL or platelet count < 100 x 10^9/L
  * Massive or rapidly progressive splenomegaly (> 6 cm below left costal margin)
  * Massive (> 10 cm) or rapidly progressive lymphadenopathy
* Life expectancy >= 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) unless due to Gilbert's disease; if total bilirubin is > 1.5 x ULN, a direct bilirubin should be performed and must be < 1.5 mg/dL for Gilbert's to be diagnosed
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 ULN
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 times ULN
* Creatinine =< 1.5 times ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x ULN
* A non-transfused platelet count >= 30 x 10^9/L
* Neutrophil count (absolute neutrophil count [ANC]) >= 1 x 10^9/L
* Hemoglobin (Hgb) >= 8 g/dL
* Note: cytopenias due to bone marrow failure are common in patients with relapsed CLL requiring treatment; accordingly, normal bone marrow function is NOT required for participation
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete patient diaries and questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to return to North Central Cancer Treatment Group (NCCTG) enrolling institution for follow-up
* Willing to provide blood samples for correlative research purposes
* Willing to provide bone marrow aspirate (body fluid) for correlative research purposes
* MAYO ROCHESTER ONLY: willing to provide bone marrow core biopsy tissue for correlative research purposes
* Willing to provide bone marrow biopsy for central pathology review (all patients)
* Able to swallow whole tablets; NOTE: nasogastric or gastrostomy (G) tube administration is not allowed; tablets must not be crushed or chewed

Exclusion Criteria:

* Prior treatment with bendamustine
* Prior treatment with any experimental Akt inhibitors
* More than 2 previous purine nucleoside based-therapy (i.e. fludarabine, pentostatin, or cladribine)
* More than 2 previous alkylating agent based-therapy (i.e. cyclophosphamide, chlorambucil)
* More than 3 total prior lines of therapy for CLL
* Primary refractory disease as defined by progression while receiving or within 6 months of completion of a chemoimmunotherapy regimen such as fludarabine, cyclophosphamide and rituximab (FCR) or pentostatin, cyclophosphamide and rituximab (PCR)
* PHASE II ONLY: FISH abnormality of 17P deletions; (note: patients with 17P deletions will be included in Phase I but will be excluded in Phase II unless enough activity is found in the Phase I)
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens; including but not limited to the following:

  * New York Heart Association class III or IV heart disease
  * Recent myocardial infarction (< 1 month)
  * Uncontrolled infection
  * Known infection with the human immunodeficiency virus (HIV/acquired immune deficiency syndrome [AIDS]) and/or patients taking highly active antiretroviral therapy (HAART) as further severe immunosuppression with this regimen may occur
  * Infection with known chronic, active hepatitis C
  * Positive serology for hepatitis B (HB) defined as a positive test for hepatitis B surface antigen (HBsAg); in addition, if negative for HBsAg but hepatitis B core antibody (HBcAb) positive (regardless of hepatitis B surface antibody [HBsAb] status), a HB deoxyribonucleic acid (DNA) test will be performed and if positive the subject will be excluded
  * Uncontrolled diabetes defined as hemoglobin A1c (HbA1c) >= 8 or fasting blood glucose >= 140 mg/dL
* Any of the following:

  * History of significant ventricular arrhythmia in the last 5 years including: ventricular tachycardia or ventricular fibrillation
  * Corrected QT (QTc) prolongation on baseline electrocardiogram (ECG) (defined as a QTc interval > 450 msec for males and QTc interval > 470 msec for females)
  * Currently using a medication known to cause prolonged QTc which cannot be discontinued; note: other medications with possible risk of prolonged QTc are allowed but should be used with caution; patients using these medications should be monitored accordingly
  * Ventricular arrhythmia on baseline ECG (ventricular tachycardia or ventricular fibrillation >= 3 beats in a row)
  * Second or third degree heart block
* Receiving any other investigational agent concurrently which would be considered as a treatment for the primary neoplasm
* Other active primary malignancy requiring treatment or which limits survival to < 24 months
* Any major surgery =< 28 days prior to registration
* Any radiation therapy =< 4 weeks prior to registration
* Current use of corticosteroids; EXCEPTION: low doses of steroids (< 10 mg of prednisone or equivalent dose of other steroid) used for treatment of non-hematologic medical conditions; NOTE: previous use of corticosteroids is allowed
* Active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment; NOTE: patients who have a positive Coombs test but no evidence of hemolysis are NOT excluded from participation
* Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450 3A4 (CYP450 3A4); use of the following strong or moderate inhibitors are prohibited =< 7 days prior to registration:

  * Strong inhibitors of CYP3A4

    * Indinavir
    * Nelfinavir
    * Ritonavir
    * Clarithromycin
    * Itraconazole
    * Ketoconazole
    * Nefazodone
    * Saquinavir
    * Telithromycin
  * Moderate inhibitors of CYP3A4

    * Aprepitant
    * Erythromycin
    * Fluconazole
    * Grapefruit juice
    * Verapamil
    * Diltiazem
* Receiving any medications or substances that are inducers of CYP450 3A4; use of the following inducers is prohibited =< 12 days prior to registration

  * Inducers of CYP3A4

    * Efavirenz
    * Nevirapine
    * Carbamazepine
    * Modafinil
    * Phenobarbital
    * Phenytoin
    * Pioglitazone
    * Rifabutin
    * Rifampin
    * St. John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Ding, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (44):
- United States (44):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 1: Patients receive:
  Cycle 1:
  1. Akt inhibitor MK2206 PO 90 mg on days 1, 8, 15, and 22 (days 1, 8, 15, 22)
  2. Rituximab IV 375 mg/m^2 on day 8.
  3. Bendamustine IV 70 mg/m^2 on day 8 and 9.
  Cycles 2-6:
  1. Akt inhibitor MK2206 PO on days 1, 8, 15, and 22 (days 1, 8, 15, 22, and 29)
  2. Rituximab IV 500 mg/m^2 on day 1.
  3. Bendamustine IV 70 mg/m^2 on day 1 and 2.
- Phase I: Dose Level 2: Patients receive:
  Cycle 1:
  1. Akt inhibitor MK2206 PO 135 mg on days 1, 8, 15, and 22 (days 1, 8, 15, 22)
  2. Rituximab IV 375 mg/m^2 on day 8.
  3. Bendamustine IV 70 mg/m^2 on day 8 and 9.
  Cycles 2-6:
  1. Akt inhibitor MK2206 PO on days 1, 8, 15, and 22 (days 1, 8, 15, 22, and 29)
  2. Rituximab IV 500 mg/m^2 on day 1.
  3. Bendamustine IV 70 mg/m^2 on day 1 and 2.
- Phase II: Patients receive:
  Cycle 1:
  1. Akt inhibitor MK2206 PO 90 mg on days 1, 8, 15, and 22 (days 1, 8, 15, 22)
  2. Rituximab IV 375 mg/m^2 on day 8.
  3. Bendamustine IV 70 mg/m^2 on day 8 and 9.
  Cycles 2-6:
  1. Akt inhibitor MK2206 PO 90 mg on days 1, 8, 15, and 22 (days 1, 8, 15, 22, and 29)
  2. Rituximab IV 500 mg/m^2 on day 1.
  3. Bendamustine IV 70 mg/m^2 on day 1 and 2.
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Started | 6 | 4 | 5
Completed | 6 | 3 | 4
Not Completed | 0 | 1 | 1
Not completed — Ineligible prior to treatment | 0 | 0 | 1
Not completed — Ineligible after receiving treatment | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients that began protocol treatment were included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II | Total
Number analyzed (Participants) | 6 | 4 | 4 | 14
Age, Continuous [Median (Full Range); unit: years] | 67.5 [44 to 74] | 66.5 [61 to 71] | 65 [54 to 75] | 67 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 5 | 3 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Participants With Dose-Limiting Toxicity Events (Phase I)
Description: The Maximum Tolerated Dose (MTD) is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Dose-limiting toxicities include non-hematologic events graded 3 or higher and deemed at least possibly related to treatment. A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD.The number of patients reporting a dose-limiting event are reported.
Time Frame: Up to 35 days
Population: Only the patients registered to the Phase I portion of this study were analyzed for this endpoint. One of the 4 patients accrued to dose level 2 was not eligible for this endpoint. Therefore, 6 patients at Dose Level 1 and 3 patients at Dose Level 2 are included in this endpoint.
Measure: Number; unit: Patients reporting Dose-Limiting Events
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Number analyzed (Participants) | 6 | 3 | 0
Patients reporting Dose-Limiting Events | 1 | 2 |

2. Primary Outcome: Proportion of Complete Response Defined to be a CR or CRi Noted as the Objective Status (Phase II)
Description: A Complete Response (CR) is defined by the NCI Working Group criteria and requires all of the following for a period of at least 2 months:
  * Absence of lymphadenopathy (e.g. lymph nodes >1.5 cm) by physical examination.
  * No hepatomegaly or splenomegaly by physical examination.
  * Absence of constitutional symptoms.
  * Neutrophils ≥1500/ul.
  * Platelets >100,000/ul (untransfused).
  * Hemoglobin >11.0 gm/dl (untransfused)
  * Peripheral blood lymphocytes <4000/uL
  Patients who fulfill all criteria for a CR but who have a persistent anemia, thrombocytopenia, or neutropenia related to drug toxicity rather than residual CLL will be classified as CR with incomplete marrow recovery (CRi).
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: From registration to response, up to 84 days
Population: All eligible patients treated at Dose Level 1 were included in the Phase II primary endpoint. All 6 patients from Phase I, Dose level 1 and 4 of the 5 patients registered to the Phase II portion of the study were eligible for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Level 1: Patients receive:
  Cycle 1:
  1. Akt inhibitor MK2206 PO 90 mg on days 1, 8, 15, and 22 (days 1, 8, 15, 22)
  2. Rituximab IV 375 mg/m^2 on day 8.
  3. Bendamustine IV 70 mg/m^2 on day 8 and 9.
  Cycles 2-6:
  1. Akt inhibitor MK2206 PO on days 1, 8, 15, and 22 (days 1, 8, 15, 22, and 29)
  2. Rituximab IV 500 mg/m^2 on day 1.
  3. Bendamustine IV 70 mg/m^2 on day 1 and 2.
Arm/Group | Dose Level 1
Number analyzed (Participants) | 10
percentage of participants | 50 [19 to 81]

3. Secondary Outcome: Biomarker Analysis (IgVH Gene Mutation)
Description: IgVH gene mutationwill be evaluated pre-treatment. This factors will be summarized and used to help characterize the types of patients accrued to this trial.
Time Frame: Baseline
Population: All patients that started treatment and had baseline biomarkers completed were included in this analysis. One of the 4 patients accrued to dose level 2 was not eligible for this endpoint. Therefore, 6 patients at Dose Level 1 and 3 patients at Dose Level 2 and 4 patients accrued to the Phase II portion of the study are included in this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Number analyzed (Participants) | 6 | 3 | 4
Participants
  Mutated | 0 | 0 | 1
  Unmutated | 5 | 3 | 1
  Not Done | 1 | 0 | 2

4. Secondary Outcome: Biomarker Analysis (CD38, CD49d, and ZAP-70)
Description: CD38, CD49d, and ZAP-70 status will be evaluated pre-treatment. These factors will be summarized and used to help characterize the types of patients accrued to this trial.
Time Frame: Baseline
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Number analyzed (Participants) | 6 | 3 | 4
Participants
  CD38: Positive | 4 | 1 | 1
  CD38: Negative | 2 | 2 | 3
  CD38: Not Done | 0 | 0 | 0
  CD49d: Positive | 1 | 0 | 3
  CD49d: Negative | 1 | 3 | 0
  CD49d: Not Done | 4 | 0 | 1
  ZAP-70: Positive | 6 | 1 | 1
  ZAP-70: Negative | 0 | 2 | 1
  ZAP-70: Not Done | 0 | 0 | 2

5. Secondary Outcome: Fluorescent in Situ Hybridization (FISH) Biomarker Analysis
Description: Fluorescent in situ hybridization (FISH) is a molecular cytogenetic technique that uses fluorescent probes that bind to only those parts of the chromosome with a high degree of sequence complementarity. It was developed by biomedical researchers in the early 1980s and is used to detect and localize the presence or absence of specific DNA sequences on chromosomes. In this disease group, there are recognized patterns of DNA sequences that play a role in prognostic outcomes. Patterns named 11q-, 13q-, Trisomy 12 may lead to different responses to treatments. Here we report the number of patients with each FISH prognosis evaluated pre-treatment. These factors will be summarized and used to help characterize the types of patients accrued to this trial.
Time Frame: Baseline
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Number analyzed (Participants) | 6 | 3 | 4
Participants
  11q- | 1 | 3 | 0
  Trisomy 12 | 1 | 0 | 1
  13q- | 2 | 0 | 1
  Other | 0 | 0 | 2
  Normal | 2 | 0 | 0

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved a clinical response as the date at which the patient's objective status is first noted to be a CR, CRi, CCR, nPR, or PR to the earliest date progression is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: Median follow-up of 39 months and maximum follow-up of 54 months
Population: 12 patients achieved a response and were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Patients: Patients receive:
  Cycle 1:
  1. Akt inhibitor MK2206 PO (90 or 135 mg) on days 1, 8, 15, and 22 (days 1, 8, 15, 22)
  2. Rituximab IV 375 mg/m^2 on day 8.
  3. Bendamustine IV 70 mg/m^2 on day 8 and 9.
  Cycles 2-6:
  1. Akt inhibitor MK2206 PO on days 1, 8, 15, and 22 (days 1, 8, 15, 22, and 29)
  2. Rituximab IV 500 mg/m^2 on day 1.
  3. Bendamustine IV 70 mg/m^2 on day 1 and 2.
Arm/Group | All Patients
Number analyzed (Participants) | 12
months | NA [3 to NA] — Too few events have occurred to provide a median and upper-level confidence interval.

7. Secondary Outcome: Minimal-residual Disease
Description: Minimal residual disease (MRD) will be evaluated after treatment in patients who achieve a complete clinical response. Flow cytometry will be used to detect approximately 1 CLL cell per 10,000 leukocytes following induction. A score of positive means CLL cells were found and a negative score means no CLL cells were found. The number of patients with an MRD negative score are reported here.
Time Frame: Cycle 6 assessment (maximum of 231 days post-registration)
Population: 5 patients achieved a complete response and were analyzed for MRD
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 5
Participants | 2

8. Secondary Outcome: Overall Response Rate
Description: The Overall response rate is estimated by the total number of complete or partial responses (CR, CRi, CCR, nPR, or PR) divided by the total number of evaluate patients. Complete and partial responses were scored using the NCI Working Group criteria. A Complete Response (CR, CRi, and CCR) is characterized by an absence of lymphadenopathy, heptomegaly and splenomegaly with or without normalized blood counts and bone marrow assessment . A PR is defined as having >50% decrease in lymphocyte count and reduction in sum of the products of measured nodes and an improvement in blood counts. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Time Frame: 3 months post-treatment
Population: All patients that were treated and evaluable for response were included together in this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | All Patients
Number analyzed (Participants) | 13
proportion of patients | 0.92 [0.64 to 0.998]

9. Secondary Outcome: Treatment-free Survival
Description: Treatment free survival is defined to be the time from registration to the date of initation of subsequent therapy or death. The distribution of treatment free survival will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the date of initiation of subsequent therapy or death, median follow-up time is 37 months
Population: All patients that were treated and evaluable were included in this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 13
months | 24.5 [11.3 to 50.6]

ADVERSE EVENTS:
Description: Adverse Events assessments took place at the end of each cycle during treatment. For each event, we are reporting the number of patients that reported the event. The total number of events reported will be defined as the total number of cycles in which the event was reported, not necessarily the number of independent events.
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/4 | 2/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 1 (N=6) | Phase I: Dose Level 2 (N=4) | Phase II (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 1 (N=6) | Phase I: Dose Level 2 (N=4) | Phase II (N=4)
Anemia (Blood and lymphatic system disorders) | 4 (16) | 4 (21) | 3 (19)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (5) | 0 (0) | 2 (9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (5) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (6) | 3 (8) | 2 (6)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (3) | 2 (4)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 2 (8)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (9) | 4 (10)
Platelet count decreased (Investigations) | 2 (16) | 4 (19) | 4 (26)
White blood cell decreased (Investigations) | 1 (1) | 3 (4) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (15) | 1 (7) | 3 (21)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (9) | 3 (7) | 3 (4)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less